CLINICAL TRIAL: NCT05817890
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-CYC065 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Absorption, Metabolism, and Excretion of CYC065 in Healthy Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-902
Record Dates: First submitted 2023-03-02; First posted 2023-04-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — CYC065

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Up to 8 subjects will be enrolled and studied as a single group (Experimental): The purpose of this study is to determine the absorption, metabolism, and excretion (AME) of [14C]CYC065 and to characterize and determine, where possible, the metabolites present in plasma, urine, and feces in healthy male subjects following a single oral administration.
  Interventions: Drug: Fadraciclib

INTERVENTIONS:
Drug: Fadraciclib — Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-CYC065 Following a Single Oral Dose in Healthy Male Subjects
  Other Names: CYC065

SUMMARY:
This will be a Phase 1, open-label, single dose study of the Absorption, Metabolism, and Excretion of CYC065 in healthy male subjects.

DETAILED DESCRIPTION:
Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Subjects will be admitted into the study site on Day -1 and be confined to the study site until at least Day 8 (168 hours post dose). On Day 1, subjects will receive a single oral dose of [14C]-CYC065. Subjects will be discharged if the following discharge criteria are met: plasma radioactivity levels below the limit of quantitation for 2 consecutive collections, ≥90% mass balance recovery, and ≤1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 2 consecutive 24-hour periods. If discharge criteria are not met by Day 8, subjects will remain in the study site until all discharge criteria are met up to a maximum of Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 55 years of age, inclusive.
2. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, with a total body weight ≥50 kg.
3. In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations at screening and check-in and from the physical examination at check-in, as assessed by the investigator (or designee).
4. Males will agree to use contraception.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
6. History of a minimum of 1 bowel movement per day.

Exclusion Criteria

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Confirmed (eg, 2 consecutive measurements) systolic blood pressure >140 mmHg or <90 mmHg, diastolic blood pressure >90 mmHg or <50 mmHg, and pulse rate >100 beats per minute or <40 beats per minute.
5. Positive hepatitis panel and/or positive human immunodeficiency virus test.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
The routes, rates of elimination, and mass balance | Up to Day 15
  Total radioactivity from [14C]-CYC065 recovery (fet1t2) in urine and feces
AUC for CYC065 in plasma | Up to Day 15
  To characterize the PK of CYC065 and total radioactivity following administration of [14C]CYC065 to healthy subjects
Cmax for CYC065 in plasma | Up to Day 15
  To characterize the PK of CYC065 and total radioactivity following administration of [14C]CYC065 to healthy subjects
Tmax for CYC065 in plasma | Up to Day 15
  To characterize the PK of CYC065 and total radioactivity following administration of [14C]CYC065 to healthy subjects
t½ for CYC065 in plasma | Up to Day 15
  To characterize the PK of CYC065 and total radioactivity following administration of [14C]CYC065 to healthy subjects

SECONDARY OUTCOMES:
Concentration of CYC065 metabolites | Up to Day 15
  To determine, where possible, the quantitative metabolite profiles in plasma, urine, and feces after [14C]CYC065
Incidence and severity of AEs | Up to Day 15
  To assess the safety and tolerability of [14C]CYC065 when administered to healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No